CLINICAL TRIAL: NCT03444649
Title: Epacadostat With Idarubicin and Cytarabine (EIC) for First-line Treatment of AML Patients Fit for Intensive Chemotherapy; a Phase I Study
Brief Title: Epacadostat, Idarubicin and Cytarabine (EIC) in AML
Acronym: EIC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: IMP will not be further developed
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EIC-trial
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: AML
Keywords: AML; Epacadostat; Idarubicin; Cytarabine
MeSH Terms: interventions — epacadostat; Idarubicin; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dosis finding (Experimental): Epacadostat is given for 2 cycles of 28 days at a dose according to the titration design together with Standard chemotherapy (Idarubicin and Cytarabine)
  Interventions: Drug: Epacadostat; Drug: Idarubicin; Drug: Cytarabine; Drug: Daunorubicin

INTERVENTIONS:
Drug: Epacadostat — Epacadostat orally two times daily (BID) for two cycles (28 days each) in combination with standard induction chemotherapy (Idarubicin and Cytarabine)
Drug: Idarubicin — Standard chemotherapy d1-d3 cycle 1
Drug: Cytarabine — Standard chemotherapy d1-d7 cycle 1 and 2
Drug: Daunorubicin — Standard chemotherapy d1-3 cycle 2

SUMMARY:
This trial assess the maximum tolerated dose (MTD) and to characterize dose-limiting toxicities (DLTs) of epacadostat when added to the anthracycline/cytarabine combination as first-line induction treatment in AML patients fit for intensive treatment

DETAILED DESCRIPTION:
Background and Rationale:

Epacadostat (INCB024360) is an Inhibitor of Indoleamine 2,3- dioxygenase 1 (IDO1). Indoleamine 2,3- dioxygenase 1 (IDO1) is a 403 amino acid cytosolic haem enzyme encoded by the INDO gene on human chromosome 8p22. IDO1 is responsible for the catabolism of the essential amino acid tryptophan (trp) to kynurenine (kyn) within immune cells and a subset of tumor cells resulting in inhibition of antitumor cell-mediated immune responses. Increased IDO activity correlates with lower CR rates and shorter OS in AML.

Objective:

The primary objective is to determine the maximum tolerated dose (MTD) and to characterize dose-limiting toxicities (DLTs) of epacadostat when added to the anthracycline/cytarabine combination as first-line induction treatment in AML patients fit for intensive Treatment.

Study Duration:

Phase I part will last from 3 to 18 months (permitting the enrolment of minimum of 3 and a maximum of 18 patients).

ELIGIBILITY:
Inclusion Criteria:

* AML (according to the 2016 World Health Organization (WHO) classification definition of ≥ 20% blasts; Arber et al, 2016) suitable for intensive treatment (including stem cell transplantation) with a curative intent.
* Patients must be aged > 18 years, and must have given voluntary written informed consent.
* Women of childbearing potential having a negative serum pregnancy test at screening or at least within 48 hours before start with epacadostat, and willing to use an effective contraceptive method (intrauterine devices, hormonal contraceptives, contraceptive pill, implants, transdermal patches, hormonal vaginal devices, infusions with prolonged release) during the study and for at least 6 months after the last study drug administration
* Men willing to use an effective contraceptive method (eg, condom, vasectomy) during the study and for at least 6 months after the last study drug administration.

Exclusion Criteria:

* Prior or concurrent malignancy, except for the following: adequately treated basal cell or squamous cell skin cancer, or any other cancer from which the subject has been disease-free for more than 6 months.
* Any previous AML or MDS chemotherapy (with the exception of hydroxyurea/Litalir® for leukocyte control which should be discontinued by the first day of induction chemotherapy
* Treatment with any investigational product within 4 weeks before the first administration of epacadostat (INCB024360)
* Abnormal organ function if not caused by the underlying disease as considered by the treating physician
* Use of immune-suppressive agents for the past 4 weeks before the first administration of epacadostat (INCB024360). For regular use of systemic corticosteroids, subjects may only be included after stepwise discontinuation to be free of steroids for a minimum of 5 days before the first administration of epacadostat (INCB024360)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Dose finding | 30 days
  To determine the maximum tolerated dose (MTD) and to characterize dose-limiting toxicities (DLTs) of epacadostat

SECONDARY OUTCOMES:
Rate of morphologic complete remission (CR) | 60 days
  Bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count > 1.0G/L (1000/μL); platelet count > 100 x G/L (100.000/μL); independence of red cell transfusions.
Adverse events | 90 days
  Number of patients experiencing toxicity (Adverse Events)
Overall survival | 12 months
  Number of patients alive after 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Medical Oncology, University Hospital Berne, Bern, Switzerland